CLINICAL TRIAL: NCT06493227
Title: The Practice of Routine Extended Perioperative Administration of Fibrinolysis Inhibitors to Reduce the Risk of Bleeding in Cardiac Surgery. Multicenter Prospective Randomized Cluster Crossover Study
Brief Title: Extended Perioperative Administration of Fibrinolysis Inhibitors After Cardiac Surgery
Acronym: PRIORITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Deputy Director for Science, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRIORITY
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Thoracic Surgery; Heart Diseases; Fibrinolysis Shutdown
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraoperative strategy (Active Comparator): Policy of no routine use of fibrinolysis inhibitors after surgery. Patients in this group will receive the center's routine prophylactic dose of fibrinolysis inhibitor, which is 100%, during surgery.
  Interventions: Other: No routine fibrinolysis inhibitors after surgery
- Intraoperative and postoperative strategy (Experimental): Policy of routine use of fibrinolysis inhibitors 4 hours after surgery. Patients in this group will receive 70% of the routine prophylactic dose of fibrinolysis inhibitor administered by the center during surgery. Additionally, they will receive 30% of the dose as an IV infusion within 4 hours after the surgery.
  Interventions: Other: Routine fibrinolysis inhibitors after surgery

INTERVENTIONS:
Other: No routine fibrinolysis inhibitors after surgery — Tranexamic acid or epsilon-aminocaproic acid should be administered intravenously during surgery. The dosage and method of administration should be followed according to the routine practice of the participating site.
  Arms: Intraoperative strategy
Other: Routine fibrinolysis inhibitors after surgery — During surgery, it is recommended to administer 70% of the routine dose of Tranexamic acid or epsilon-aminocaproic acid intravenously. Following the surgery, the remaining 30% of this dose should be administered as a continuous intravenous infusion over the course of the first 4 hours.
  Arms: Intraoperative and postoperative strategy

SUMMARY:
PRIORITY is a pragmatic, multi-center, cluster crossover trial that aims to evaluate whether implementing a policy of routine extended (intraoperative and 4 hour after transfer to ICU) use of fibrinolysis inhibitors leads to a decrease in post-operative blood transfusion compared to a policy that only involves intraoperative use.

DETAILED DESCRIPTION:
Routine use of fibrinolysis inhibitors is strongly recommended in cardiac surgery (recommendation level 1A). However, despite numerous studies on the pharmacodynamics and clinical effects of these drugs, there is still no consensus on the optimal dose and dosage regimen. As a result, there is wide variability in the use of fibrinolysis inhibitors across different clinics. Several studies have shown that peak activation of fibrinolysis occurs during cardiopulmonary bypass. However, elevated levels of markers of fibrinolytic activity in the blood plasma are observed for at least 2 hours after surgery and 4 hours after heparin neutralization. This suggests the potential for extended use of fibrinolysis inhibitors after surgery. There have been limited attempts to investigate the effectiveness of postoperative administration of fibrinolysis inhibitors, and these studies have been conducted on small samples or with retrospective designs. The authors of these studies were unable to identify the benefits of postoperative administration in terms of reducing bleeding risk and the need for blood transfusions. However, postoperative infusion of fibrinolysis inhibitors demonstrated a comparable safety profile. There is evidence suggesting that repeated administration of fibrinolysis inhibitors after cardiopulmonary bypass, rather than a single dose at the beginning of surgery, may be more beneficial. Due to uncertainty regarding the best approach (routine extended use of fibrinolysis inhibitors or no routine extended use of fibrinolysis inhibitors), we will compare the effects of a hospital policy that includes routine administration of fibrinolysis inhibitors 4 hours after surgery to a policy that avoids routine postoperative administration. The comparison will focus on the blood transfusion requirement during hospitalization among patients undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. A hospital that performs a minimum of 250 open heart interventions per year.
2. Consent from hospital physicians regarding the prophylactic use of fibrinolysis inhibitors (more than 95% of physicians involved in the treatment of adult patients (>18 years) agree to adhere to the strategy of using fibrinolysis inhibitors as prescribed by the study protocol).

Exclusion Criteria:

* Hospital does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1373 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
RBC transfusion | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  The rate of red blood cells transfusion during the hospitalisation.

SECONDARY OUTCOMES:
Hospital stay | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Duration of stay in the hospital, days
Redo surgery requirement | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Rate of reexplorations during the initial hospitalisation
Haemoglobin on discharge | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  The last available blood haemoglobin level before the discharge
Total blood products requirement | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Number blood products transfused, units

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Cardiac surgery department, Saint-Petersburg state university hospital, Saint Petersburg
  - St. Petersburg State University Hospital, Saint Petersburg